CLINICAL TRIAL: NCT04979845
Title: The Effect on Telerehabilitation on Fatigue and Sleep Quality in Patients With Multiple Sclerosis
Brief Title: Telerehabilitation in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021.808
Record Dates: First submitted 2021-07-27; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation; Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental)
  Interventions: Other: Telerehabilitation
- Video exercise (Active Comparator)
  Interventions: Other: Video exercise

INTERVENTIONS:
Other: Telerehabilitation — Patients will receive telerehabilitation sessions for 12 weeks including aerobic and strengthening exercises
  Arms: Telerehabilitation
Other: Video exercise — Patients will receive video instructions for home based exercises
  Arms: Video exercise

SUMMARY:
Patients with multiple sclerosis will be randomized into two groups. One group will receive live telerehabilitation sessions 3 times a week over a course of three months. The other group will receive video instructions for aerobic and strengthening exercises. Patients fatigue, sleep quality and quality of life will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple scleroisis

Exclusion Criteria:

* Any musculoskeletal condition preventing patients to actively participate in exercise sessions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Scale | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaya A, Karadag-Saygi E, Kucukosmanoglu Z, Kenis-Coskun O, Agan Yildirim K. Effect of Telerehabilitation Exercise Program on Sleep Quality and Fatigue in Individuals With Multiple Sclerosis. Ann Rehabil Med. 2025 Oct;49(5):302-309. doi: 10.5535/arm.250010. Epub 2025 Oct 31. PMID 41177152